CLINICAL TRIAL: NCT07052565
Title: An Exploratory Clinical Study of Enhanced Autologous CAR-T Cell Injection (ECAR01) Targeting BCMA and CD19 in the Treatment of Refractory Autoimmune Diseases
Brief Title: CAR-T Cells Therapy for Patients With Autoimmune Diseases
Acronym: ECAR01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWKCART24101501
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Autoimmune Diseases
Keywords: systemic sclerosis; dry syndrome; rheumatoid arthritis; systemic lupus erythematosus
MeSH Terms: conditions — Autoimmune Diseases; Scleroderma, Systemic; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-BCMA and CD19 CART (Experimental): Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CART infusion. A dose of Anti-BCMA and CD19 CART will be infused on day 0.
  Interventions: Drug: Anti-BCMA and CD19 CART cells will be injected intravenously on a one-time basis

INTERVENTIONS:
Drug: Anti-BCMA and CD19 CART cells will be injected intravenously on a one-time basis — A single intravenous infusion of anti-BCMA and CD19 CART cells (dose-escalating infusion of 1.0-6.0 x10^5 CART cells/kg）

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with refractory autoimmune diseases. This study aims to evaluate the safety and efficacy of the treatment with Anti-BCMA and CD19 CART

DETAILED DESCRIPTION:
This study is a single-center, single-arm, non-blinded, 3+3 dose-escalation designed investigator initiated trial study, evaluating the safety, efficacy, and therapeutic assessment of ECAR01 injection in patients with refractory autoimmune diseases. The specific research protocol can be adjusted by the researchers based on the patient's condition. Patients with refractory autoimmune diseases who meet the inclusion and exclusion criteria are included. After peripheral blood collection and chemotherapy pretreatment, the subjects undergo CAR-T cell infusion. The three dose groups are the low-dose group (1×10^5/kg, number of CAR-T cells per kg of subject's weight, the same below), the medium-dose group (3×10^5/kg), and the high-dose group (6×10^5/kg). Clinicians can also adjust the drug dose based on actual conditions. Given the particularity of cell preparation doses, each dose group allows for a ±20% fluctuation in the actual drug dose.

ELIGIBILITY:
Inclusion Criteria:

* ( 1) At the time of signing the informed consent form, be at least 18 years of age, both male and female.

  (2) Bone marrow hematopoietic function satisfies: white blood cell count≥3×10^9/L; Centrocyte count ≥1×10^9/L (no colony-stimulating factor received within 2 weeks prior to screening); Hemoglobin ≥ 60g/L.

  (3)ALT≤3×ULN; AST≤3×ULN； TBIL≤3×ULN。 (4) Renal function satisfaction: creatinine clearance CrCl≥30mL/min. (5) INR≤1.5×ULN , PT≤1.5×ULN. (6)RA:Documented diagnosis of RA which fulfills the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria ; 3 months after use of 1 or more csDMARDs and 1 or more bDMARDs prior to screening: 1) DAS28-ESR>3.2 or CDAI>10; or 2) the dose of the hormone (prednisone or equivalent) cannot be reduced to less than 7.5 mg/day; or 3) the number of swollen and/or tender joints ≥3; Treatment with stable 1 or more cs DMARD(s) and/or bDMARDs prior to enrollment as follows: methotrexate for at least 12 weeks and at a dose of 7.5-25mg/week for at least 4 weeks; Stable use of hydroxychloroquine dose ≤ 400 mg/day for at least 4 weeks; Stable oral sulfasalazine for at least 4 weeks 1~3 g/d; Stable oral leflunomide 10-20 mg/day for at least 4 weeks.

  (7)systemic lupus erythematosus : Diagnosis of systemic lupus erythematosus according to the SLE classification criteria of the 2019 EULAR/ACR; History of systemic lupus erythematosus for at least 6 months prior to screening and active disease for 2 months after use of standard treatment regimens prior to screening; BILAG-2004 assesses the presence of at least 1 Grade A or 2 Grade B organ scores; Positive antinuclear antibody, or positive anti-ds-DNA antibody, or positive anti-Sm antibody; SLEDAI-2000 score ≥8 during the screening period.

  (8)Sjögren's syndrome : Diagnosis of Sjögren's syndrome according to the 2002 International Classification of Primary Sjögren's Syndrome or the 2016 ACR/EULAR classification criteria; Diagnosed with pSS-TP and platelet count < 30×10^9/L; Sjögren's syndrome Disease Activity Index (ESSDAI) score ≥5 during the screening period; Sjögren's syndrome for at least 6 months prior to screening and active disease 2 months after use of conventional treatment regimens prior to screening. Use of immunomodulatory drugs for more than 6 months.

  (9)systemic sclerosis : Diagnosis of systemic sclerosis according to the 2013 ACR classification criteria for systemic sclerosis. Positive antinuclear antibody at screening. Presence of clear evidence of HRCT progression. History of systemic sclerosis prior to screening for at least 6 months and active disease for 2 months after use of conventional treatment regimens prior to screening.

Exclusion Criteria:

* (1) Clinically significant central nervous system diseases or pathological changes not caused by the disease itself before screening, including but not limited to: stroke, stroke, aneurysm, epilepsy, convulsions, aphasia, severe head injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome or mental disorder.(2) Those with relatively serious heart disease, such as angina, myocardial infarction, heart failure and arrhythmia.(3) History of major organ transplantation or hematopoietic stem cell/bone marrow transplantation.(4) Vaccination, B-cell targeted therapy within 4 weeks prior to screening.(5) History of any malignant neoplastic disease.(6) Patients with end-stage renal failure.(7) The presence or suspicion of uncontrollable fungal, bacterial, viral, or other infections.(8) History of severe allergy to drugs used in clinical studies or raw and excipient materials of experimental drugs, such as cyclophosphamide, fludarabine, DMSO, etc.(9) Patient has active HBV infection or HCV antibody positivity or HIV antibody positivity or syphilis positivity or CMV DNA positivity or EBV DNA positivity.(10) Pregnant or lactating females, or planning to become pregnant within 2 years after reinfusion of the trial drug; The partner of the male patient plans to become pregnant within 2 years of receiving the trial drug.(11) Evidence of active tuberculosis infection.(12) Other conditions assessed by the investigator as unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 1 years
  Total number, incidence and severity of adverse events (AEs) in patients of SCAR02 infusion. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.

SECONDARY OUTCOMES:
The change of CAR copy number in peripheral blood was investigated by comparison with baseline | up to 1 years
  Peripheral blood CAR copy concentrations (copies/µL) will be detected using QPCR
Disease activity was assessed by DAS28 | up to 1 years
  DAS28 was used to assess disease activity, and the number of swelling and tenderness in 28 joints was examined, Min/Max Value: Not specified,with higher scores representing worse disease status.
Modified Rodnan Skin Score assesses disease activity in patients | up to 1 years
  Disease activity was assessed by Modified Rodnan Skin Score Modified Rodnan Skin Score: The modified Rodnan Skin Score was used to assess the degree of skin involvement in patients with systemic sclerosis, and the thickness and hardness of the skin on the patient's head and neck, upper limbs, fingers, chest, abdomen, lower limbs, feet, etc., each part was divided into 0 (normal), 1 (mild thickening), 2 (moderate thickening), and 3 (severe thickening) according to the skin involvement, and the scores of each part were added together to obtain a total score, The higher the score, the worse the skin lesion status in patients with systemic sclerosis.
SLEDAI assesses disease activity in patients | up to 1 years
  SLEDAI was used to evaluate the disease activity of patients with systemic lupus erythematosus, and the clinical symptoms and laboratory examination indicators of the patients were quantitatively scored.The SLEDAI score ranges from 0~105 points, and the higher the score, and the higher the score, the worse the disease status of systemic lupus erythematosus.
BILAG-2004 assesses disease activity in patients | up to 1 years
  BILAG-2004 score: BILAG-2004 was used to evaluate the disease activity of patients with systemic lupus erythematosus, and the clinical manifestations of patients in 10 systemic domains were scored according to the involvement of each domain according to the five grades of A (very severe), B (moderately severe), C (mild), D (in the past, now none), and E (never), and the scores in each domain were comprehensively weighted, and the higher the score, the worse the disease status of systemic lupus erythematosus.
Change from baseline in Physician's Global Assessment of Arthritis (PGA) (VAS) | up to 1 years
  The investigator/sub-investigator assesses the participant's disease activity on a VAS of 0 - 3 mm on the physician assessment table
Change from baseline in ESR | up to 1 years
  ESR will be measured with blood samples
ACR70 response rate | up to 1 years
  The ACR70 response indicates a 70% improvement in all criteria used in the ACR70 assessment
Clinical response for Sjögren's Syndrome | up to 1 years
  Sjögren's tool for assessing response (STAR): Min/Max Value: Not specified; a decrease in score indicates improvement; higher scores indicate worse outcome
Change from baseline in participant's assessment of pain (VAS) | up to 1 years
  Using the VAS pain visual analog scale to visually display the patient's pain level, using a 10cm long scale, there are 10 scales from 0 to 10, 0 represents no pain, 10 represents severe pain, and let the patient choose a scale that meets his pain feelings
HAQ health assessment | up to 1 years
  The HAQ health assessment questionnaire was used to assess disease activity, and 8 questions of daily activities were set up for patients to answer, with each question scoring 0-3, 0 points indicating no difficulty, 1 point being somewhat difficult, 2 points being difficult or needing help, and 3 points being unable to complete. The higher the patient's score, the worse the function
Change from baseline in CRP | up to 1 years
  CRP will be measured with blood samples

CONTACTS AND LOCATIONS:
Overall Officials: wang xing bing, M.D, Principal Investigator — Anhui Provincial Hospital; chen zhu, M.D, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui Provincial Hospital, Hefei, China